CLINICAL TRIAL: NCT05053594
Title: Different Doses of Neostigmine for Reversal of Cisatracurium-induced Moderate Neuromuscular Blockade in Children Under Sevoflurane Anesthesia
Brief Title: Different Doses of Neostigmine for Reversal of Moderate Neuromuscular Blockade in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Toshiyuki Moro, Professor, Pontificia Universidade Catolica de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE 46436121.0.0000.5373
Record Dates: First submitted 2021-08-13; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Neuromuscular Blockade; Neuromuscular Block, Residual; Neuromuscular Block Prolonged
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Neostigmine

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: For each patient, an opaque envelope will be prepared, sealed and numbered sequentially containing the group to which the patient will be allocated. A list of randomized computer-generated numbers (www.random.org) will be used for this purpose. No surgeon, assistant, nurse and anesthesiologist involved in anesthesia control or data collection will be aware of the dose of neostigmine to be administered. An anesthesiologist not involved in the study will be responsible for preparing the solution containing neostigmine and atropine (diluted with saline solution until complete 10mL) according to the group to which each patient belongs. The syringes will be similar and identified only with a label with the word "reversal".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group N10 (Experimental): Reversal with neostigmine 10 mcg/kg and atropine 5 mcg/kg
  Interventions: Drug: Neostigmine 10 mcg/kg
- Group N20 (Experimental): Reversal with neostigmine 20 mcg/kg and atropine 10 mcg/kg
  Interventions: Drug: Neostigmine 20 mcg/kg
- Group N30 (Experimental): Reversal with neostigmine 30 mcg/kg and atropine 15 mcg/kg
  Interventions: Drug: Neostigmine 30 mcg/kg
- Group P (Placebo Comparator): Spontaneous reversal (placebo)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Neostigmine 10 mcg/kg — Once the third response to TOF is obtained, neostigmine 10 mcg/kg will be administered
  Arms: Group N10
Drug: Neostigmine 20 mcg/kg — Once the third response to TOF is obtained, neostigmine 20 mcg/kg will be administered
  Arms: Group N20
Drug: Neostigmine 30 mcg/kg — Once the third response to TOF is obtained, neostigmine 30 mcg/kg will be administered
  Arms: Group N30
Other: Placebo — Once the third response to TOF is obtained, saline will be administered
  Arms: Group P

SUMMARY:
There is no recent information on the required dose of neostigmine for the reversal of cisatracurium-induced moderate neuromuscular blockade (NMB) [Train-of-four (TOF) count = 1-3)] in children. The aim of this study will be to evaluate by means of a prospective, randomized and double-blinded clinical trial, the time required for reversal of moderate NMB (TOFc 3) to T4/T1 (TOF ratio, TOFr) > 0.9 and TOFr = 1.0 after administration of different doses of neostigmine (10, 20 or 30 mcg/kg) or placebo in children undergoing inhalational (sevoflurane) general anesthesia. In addition, the probability of NMB reversal in less than 10 minutes, the presence of bradycardia, respiratory complications and postoperative vomiting will be evaluated. The time for reversal is expected to be inversely proportional to the administered dose of neostigmine.

DETAILED DESCRIPTION:
Children aged between 2 and 10 years old submitted to general anesthesia to perform tonsillectomy associated or not to adenoidectomy and will be evaluated in this prospective and randomized study. Patients will be randomly distributed into one of 4 groups according to the dose of neostigmine used for NMB reversal:

* Group N10: reversal with neostigmine 10 mcg/kg and atropine 5 mcg/kg
* Group N20: reversal with neostigmine 20 mcg/kg and atropine 10 mcg/kg
* Group N30: reversal with neostigmine 30 mcg/kg and atropine 15 mcg/kg
* Group P: spontaneous reversal (placebo)

For each patient, an opaque envelope will be prepared, sealed and numbered sequentially containing the group to which the patient will be allocated. A list of randomized computer-generated numbers (www.random.org) will be used for this purpose. No surgeon, assistant nursing, and anesthesiologist involved in anesthesia control or data collection will be aware of the dose of neostigmine to be administered. An anesthesiologist not involved in the study will be responsible for preparing the solution containing neostigmine and atropine (diluted with saline solution until complete 10mL) according to the group to which each patient belongs. The syringes will be similar and identified only with a label with the word "reversal".

STUDY SEQUENCE

Anaesthesia No child will receive preanesthetic medication. After entry into the operating room, all patients will be monitored with cardioscope, noninvasive blood pressure, pulse oximetry and, after tracheal intubation, with capnography. In all children, venous access will be obtained in one of the upper limbs after induction under facial mask with sevoflurane (6%) in mixture with O2 5 L/min. After pre-oxygenation, tracheal intubation will be performed after intravenous fentanyl (3 mcg/kg) and cisatracurium (0.1 mg/kg). Anesthesia maintenance will be based on sevoflurane (1 to 2 CAM) diluted in O2/air flow (60%) 2 L/min. Ventilation will be controlled, with tidal volume and respiratory rate adjusted for the maintenance of PETCO2 between 30 and 40 mmHg. When there is a suspicion of inadequate anesthesia plan the concentration of sevoflurane will be increased and if adequacy is not sufficient, additional fentanyl bolus (1 mcg/kg) will be administered. Repeated doses of cisatracurium (0.02 mg/kg) will be used to maintain TOFc < 4. All patients will receive clonidine 2 mcg/kg intravenously, dexamethasone 0.1 mg/kg, ondansetron 0.1 mg/kg, dipyrone 30 mg/kg and morphine 0.1 mg/kg. Hydration will be performed with 0.9% saline (2 mL/kg/h). The central temperature will be kept above 36 degrees Celsius and peripheral (tenar eminence of the monitored palm) above 32 degrees Celsius. The NMB reversal will be performed when TOFc 3.

Monitoring of neuromuscular blockade NMB will be monitored by the acceleromyography method (TOF Watch ®; Schering-Plough) as recommended for use in clinical research. The acceleration transducer will be fixed on the volar side of the distal phalanx of the thumb. Venous access and blood pressure cuff will be positioned on the opposite arm to the limb used for NMB monitoring. After cleaning the skin in the path of the ulnar nerve in the forearm, the electrodes will be positioned at the height of the wrist with a distance between 3 to 6 cm between them. Calibration will be performed after automatically after a 50 Hz tetanic stimulation for 5 seconds. The stimulation (Train-of-Four, TOF) will be applied every 15 seconds for 2 minutes before cisatracurium administration. No additional doses of NMB will be given. Once the third response to TOF is obtained, a dose of neostigmine (10, 20 or 30 mcg/kg) will be administered and the time until the TOF reaches values equal to 0.9 and 1.0 will be recorded. The primary outcome will be the time required for the reversal of moderate NMB (TOFc 3) up to TOFr 0.9 and TOFr 1.0. In addition, the probability of reversal of NMB in less than 10 minutes after administration of different doses of neostigmine will be evaluated. The sample size will be based on a previous study that determined the need for 12 patients per group to detect a difference of 4 minutes and a standard deviation of 3 minutes with a power of 80% and alpha error of 5%. 9 Considering the possible losses, a total of 60 children will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Children physical status according to the American Society of Anesthesiologists I and II
* Submitted to general anesthesia to perform tonsillectomy associated or not with adenoidectomy

Exclusion Criteria:

* Refusal to participate in the study
* Presence of kidney, liver or neuromuscular disease
* Contraindication to the use of any drug used in the study
* Body mass index (BMI) ≥ 30.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
Time for complete reversal of moderate NMB | Time from neostigmine administration up 60 minutes after complete reversal
  Time required for reversal of TOFc 3 to T4/T1 (TOF ratio, TOFr) = 1.0

SECONDARY OUTCOMES:
Time for reversal of moderate NMB to TOFr 0,9 | Time from neostigmine administration up to 60 minutes after complete reversal
  Time required for reversal of TOFc 3 to T4/T1 (TOF ratio, TOFr) > 0.9
Probability of NMB reversal in less than 10 minutes | Time from neostigmine administration up to 10 minutes
  Probability of TOFc 3 to TOFr 1.0 in less than 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo T Moro, MD, Principal Investigator — Pontificia Catholic University of São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Data will be available if requested by e-mail (edumoro85@gmail.com)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From Clinical trials approval up to 12 months
Access Criteria: If requested by email